CLINICAL TRIAL: NCT07303998
Title: Feasibility and Effect of Remotely Supervised Transcranial Direct Current Stimulation With Chair Yoga for Chronic Knee Pain Management in Older Adults With Alzheimer's Disease and Related Dementias.
Brief Title: Remote tDCS and Chair Yoga for Chronic Knee Pain in Alzheimer's Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Juyoung Park, Professor, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jpark13
Record Dates: First submitted 2025-10-13; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer&Amp;#39;s Disease; Other Dementias
Keywords: transcranial direct current stimulation; chair yoga; older adults; Chronic knee pain; Dementias; online chair yoga; seniors
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active Chair Yoga paired with active tDCS (Experimental): Active Chair Yoga paired with active tDCS
  Interventions: Device: Active tDCS paired with active online chair yoga

INTERVENTIONS:
Device: Active tDCS paired with active online chair yoga — Active tDCS with a constant current of 2 milli amperes (mA) will be applied for 20 minutes daily for 1 week, and 20 minutes 3 times per week for 3 weeks via the Soterix 1x1 tDCS mini-CT Stimulator device with headgear and saline-soaked surface sponge electrodes. Online chair yoga therapy lasting 30 minutes will be conducted via Zoom by a yoga therapist immediately after each tDCS session.
  Other Names: online chair yoga; trans-direct current stimulation

SUMMARY:
This study aims to evaluate the feasibility, acceptability, and preliminary effects of a home-based, remotely supervised intervention combining transcranial direct current stimulation (tDCS) and online chair yoga (OCY) to manage chronic knee pain in older adults with Alzheimer's Disease and Related Dementias (ADRD). Chronic knee pain is prevalent among individuals with ADRD and is often underdiagnosed and undertreated, contributing to neuropsychiatric symptoms, reduced quality of life, and increased caregiver burden. Current pharmacological options, such as opioids, pose risks of adverse events in this population.

tDCS is a safe, noninvasive technique that uses low-intensity electrical current to modulate brain activity and may improve pain perception by targeting central mechanisms. Chair yoga is a mind-body intervention shown to improve pain and mood in older adults, including those with dementia. This study proposes that combining tDCS and OCY may have synergistic benefits in reducing pain and enhancing function.

Participants will include older adults aged 60+ with mild to moderate ADRD and chronic knee pain, along with their caregivers. Over four weeks, participants will complete 14 supervised sessions of combined tDCS and OCY at home. Outcomes include feasibility, satisfaction, pain intensity, pain interference, neuropsychiatric symptoms, sleep disturbance, cognitive function, mobility, and quality of life. Neurophysiological measures (e.g., fNIRS, EEG, HF-HRV) will also be assessed to explore underlying mechanisms.

This study seeks to lay the foundation for future large-scale randomized controlled trials of home-based nonpharmacological interventions for chronic pain in ADRD.

DETAILED DESCRIPTION:
Older adults with ADRD frequently experience chronic pain, particularly knee pain, which is associated with worse behavioral symptoms and faster cognitive decline. Despite its impact, pain is often inadequately treated in this population due to communication difficulties and the risks associated with pharmacological treatments, especially opioids.

Transcranial direct current stimulation (tDCS) is a promising nonpharmacological therapy that delivers low-intensity electrical current to modulate cortical excitability. Research suggests that tDCS can reduce clinical and experimental pain and improve pain processing, particularly when targeted to the motor cortex. Our group has demonstrated the safety and efficacy of home-based, remotely supervised tDCS in older adults, including those with ADRD.

Chair yoga (CY), a modified yoga intervention involving seated or chair-supported postures, is also safe and effective for older adults with chronic pain and cognitive impairment. CY has demonstrated benefits in reducing pain, improving mood, and promoting physical activity with minimal risk of falls. Evidence suggests that yoga interventions may enhance central pain modulation and reduce neuropsychiatric symptoms.

This pilot study tests a novel combination of tDCS and online CY (OCY) in a home-based setting. We hypothesize that combining tDCS and OCY will reduce chronic knee pain and improve related symptoms in older adults with ADRD.

Participants will be recruited from geriatric outpatient clinics and community settings. Eligible participants will be 60 years or older, have mild to moderate ADRD, and experience chronic knee pain. The intervention will include 14 sessions over four weeks. All sessions will be supervised remotely via a secure videoconferencing platform.

Primary outcomes are feasibility, acceptability, and satisfaction, assessed through recruitment, adherence, dropout rates, and participant feedback. Secondary outcomes include reductions in knee pain (measured by Numerical Rating Scale and MOBID-2), pain interference (PROMIS Pain Interference 4a), sleep disturbance (ActiGraph), neuropsychiatric symptoms (Neuropsychiatric Inventory Questionnaire), cognitive function (Montreal Cognitive Assessment and Cognivue), mobility (Timed Up and Go), and quality of life (QOL-AD).

Exploratory neurophysiological outcomes will include functional near-infrared spectroscopy (fNIRS) to assess pain-related brain activity, EEG for neural pain signatures, and high-frequency heart rate variability (HF-HRV) for autonomic function.

This study will help determine the feasibility and potential effects of a scalable, home-based tDCS+OCY protocol, with the goal of informing future large-scale trials and advancing personalized, nonpharmacological pain care in ADRD.

ELIGIBILITY:
Inclusion Criteria (participants):

* Live in the community (not institutionalized).
* Have a diagnosis of Alzheimer's disease and related dementias (ADRD), including Alzheimer's disease, Lewy Body Dementia, Vascular Dementia, or Multiple Etiology Dementias (MED) diagnosed by a neurologist or other healthcare provider.
* Be in mild to moderate ADRD, as indicated by a Quick Dementia Rating Scale (QDRS) score between 6 and 20.5.
* Score above 10 on the Montreal Cognitive Assessment (MoCA).
* Experience chronic knee pain (caregiver-reported average pain in the past 3 months > 40 out of 100).
* Have no planned changes to their medication regimen or other interventions for knee pain during the trial.
* Agree to participate in both transcranial direct current stimulation (tDCS) and online chair yoga (OCY).
* Be able to ambulate independently with minimal assistance (e.g., using a cane or walker) for participation in OCY and the Timed Up and Go (TUG) test. - -- Be English-speaking and able to understand verbal instructions (literacy not required).
* Be able to consent for themselves or identify a legally authorized representative who can provide written informed consent.
* Exhibit neuropsychiatric symptoms (e.g., apathy, agitation).
* Be naïve to yoga and tDCS.

Exclusion Criteria (participants):

* a history of brain surgery, brain tumor, head trauma, seizure/epilepsy, stroke, cancer affecting the head, or intracranial metal implantation;
* systemic rheumatic disorders, including rheumatoid arthritis, systemic lupus erythematosus, or fibromyalgia;
* prosthetic knee replacement or non-arthroscopic surgery to the affected knee;
* compromised skin integrity on the head in the area where electrodes will be placed;
* serious comorbidities that preclude participation in tDCS or OCY (e.g., heart failure [level IV] causing shortness of breath on exertion);
* hospitalization within the preceding year for neuropsychiatric illness that would impact knee pain or interfere with study procedures;
* use of another neurostimulation device (e.g., spinal cord stimulator, cardio-stimulator, or implanted cardioverter-defibrillator).

Inclusion Criteria (caregivers):

A caregiver is defined in this study as the person who provides care and assistance to a patient with ADRD (e.g., helping with daily activities, managing medications, ensuring safety).

* Caregivers must be at least 18 years old
* have provided care and assistance to the patient for at least 10 hours per week at the time of enrollment
* anticipate continuing to provide care and assistance for the next 4 months (until the study ends)
* be willing to receive tDCS training, administer home-based tDCS sessions, and assist the patient in attending OCY sessions
* have access to a reliable Internet connec¬tion for secure videoconferencing for real-time remote supervision
* English-speaking caregivers who can understand verbal instructions.

Exclusion Criteria (caregivers):

* alcohol/substance use disorder
* inability to understand English
* disability that would prevent assisting patients with ADRD from participating in tDCS and OCY (e.g., blindness, deafness)
* unwillingness to provide care and assistance to patients until the study is completed.
* If caregiver does not meet the inclusion/exclusion criteria, the participant will not be accepted into the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Score (NRS) of Pain | Baseline (Week 0); after each intervention session (Sessions 1-14 over Weeks 1-4); and end of intervention (Week 4).
  Clinical pain intensity will be measured by asking participants to rate their knee pain over the last 24 hours between 0 (no pain) - 10 (worst pain imaginable). The NRS has a reported Cronbach's alpha coefficient of ≥ 0.8 and is a reliable way for measuring knee pain in adults with knee osteoarthritis.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference 4a | Baseline (Week 0); after each intervention session (Sessions 1-14 over Weeks 1-4); and end of intervention (Week 4).
  The PROMIS Pain Interference 4a measures pain's impact on daily activities, with four items rated on a 5-point scale. Patients will self report this data based on their activities from the last 7 days. This tool has high reliability with a Cronbach's alpha ~0.90.
Mobilization-Observation-Behavior-Intensity-Dementia Pain Scale (MOBID-2) | Baseline (Week 0); after each intervention session (Sessions 1-14 over Weeks 1-4); and end of intervention (Week 4).
  The MOBID-2 asks caregivers to evaluates the pain of participants during specific activities(guiding hands together, turning in bed, sitting at bedside, etc.) and at specific parts of the body (head, mouth, neck, heat lungs, chest wall, etc), with a score range of 0-10; scores over 2 are clinically significant. The MOBID-2 shows high reliability with a Cronbach's alpha 0.86-0.89.
ActiGraph Watch | Continuously assessed from baseline (Week 0) through end of intervention (Week 4).
  The ActiGraph wGT3X-BT and ActiLife software objectively measures sleep disturbance. Wrist actigraphy is a valid and reliable tool for assessing sleep in patients with ADRD. Patients will be asked to wear the watch on their nondominant wrist, with caregiver assistance. Actigraphy data are analyzed to calculate sleep outcomes, including total sleep time, wake time, and daytime naps, using the standard algorithm in ActiLife software without additional hand scoring.
The Montreal Cognitive Assessment (MoCA v. 8.1) | Baseline (Week 0) and end of intervention (Week 4).
  MoCA is a 30-point test that includes 12 subtasks that cover a total of 8 cognitive domains (e.g., memory, orientation, attention/concentration, executive function), with scores ranging 0-30, with higher scores indicating better global cognitive performance. The MoCA features educational correction by the addition of 1 point for the patient with less than a 12th-grade education. The MoCA has high internal reliability (Cronbach α = .83), high test-retest reliability (ICC = 0.92), high interrater reliability (ICC = .81), and high content validity (r = .87).
Functional near-infrared spectroscopy (fNIRS) brain imaging | Baseline (Week 0) and end of intervention (Week 4).
  Pain related cortical responses will be measuring using a continuous multichannel fNIRS imaging system (LIGHTNIRS, Shimadzu, Kyoto, Japan). This instrument encompasses 8 light sources (each emitting laser light at 780, 805, and 830 nm) and 8 detectors connected to comfortable headgear using optical fibers. Optical recordings will be collected during thermal pain stimulation and punctate pain stimulation.
Heart Rate Variability Monitor | Baseline (Week 0) and end of intervention (Week 4).
  The Bittium Faros™ 180 device will be used to record continuous electrocardiogram (ECG) data for analyses of cardiac rhythms. The device samples ECG at 1000 Hz and is attached using three self-adhesive electrodes on the torso. Respiratory Sinus Arrhythmia (RSF) and Heart Rate (HR) will be measuring over 3 minutes during 3 postures (stand-sit-stand) for a total collection period of 9 minutes.
Neuropsychiatric Inventory Questionnaire (NPI-Q) | Baseline (Week 0); during intervention on Days 5, 8, 11, and 14 (Weeks 1-4); and end of intervention (Week 4).
  The NPI will be administered to the caregiver to evaluate the participant's neuropsychiatric symptomatology of dementia. The NPI uses a 4-point Likert-type scale for frequency and a 3-point Likert-type scale for severity of 12 sub-domains of dementia (e.g., delusions, hallucinations, agitation/aggression, night-time behavioral disturbances, and appetite and eating abnormalities). These are summed to yield an overall score of 0-144 (each item rated frequency X severity, totaling 0-12), with higher scores indicating greater symptoms. Internal consistency reliability of the NPI is high with a Cronbach's alpha = 0.80.
Time Up and Go Test (TUG) | Baseline (Week 0) and end of intervention (Week 4).
  TUG will measure functional mobility by timing patients as they stand from a chair, walk 10 feet, turn 180 degrees, return, and sit down. The average of three tests will be recorded in seconds. TUG is a simple and widely used tool for assessing lower limb function, mobility, and fall risk, with high inter-rater (ICC = .99) and intra-rater reliability (ICC = .99).
Cognivue Clarity | Baseline (Week 0) and end of intervention (Week 4).
  Cognivue Clarity is the first FDA-cleared computerized cognitive assessment device to evaluate a range of specific cognitive domains (e.g., motor speed, visuospatial abilities, verbal and visual episodic memory, attention, executive function, reaction time). It is an easy-to-use automated platform for evaluating and tracking cognitive impairment, with 10 separately scored subtests (2 for visuospatial functioning, 4 for perceptual processing, and 4 for memory). The 10-minute assessment provides a numerical score categorizing performance as normal, mild impairment, or moderate impairment. Classification ranges are no cognitive impairment (CI) (≥75), low-mild CI (51-74), and moderate-severe CI (≤50).
Client Satisfaction Questionnaire (CSQ-8) | End of intervention (Week 4).
  We will measure participant satisfaction with treatment using the CSQ-8. The CSQ-8 comprises eight items that are summed to yield an overall score of 8-32, with higher scores indicating greater satisfaction. The CSQ-8 has a reported Cronbach's alpha coefficient of 0.87-0.93. We will evaluate the presence and severity of possible side effects of treatment at the end of each session on a 0 (not at all) to 10 (highest degree) scale. Participants will be asked in an open-ended manner whether they experienced any side effects, and they will complete a brief questionnaire assessing side effects that can occur with tDCS or/and OCY (e.g., itching, headache, fatigue, dizziness).
Acceptability and Experience Survey | End of intervention (Week 4).
  To measure acceptability, we will administer an adapted questionnaire to patients and caregivers at the end of the intervention. Items rated from 0 (strongly disagree) to 10 (strongly agree) will include (a) ease of preparing tDCS and chair yoga props, (b) complexity and usability of the tDCS device, (c) ease of following yoga poses, (d) helpfulness of video conferences, (e) confidence in using tDCS, and (f) overall benefit of the interventions. Negative items will be reverse coded, and total scores will range from 0 to 100, with higher scores indicating greater acceptability.
Quick Dementia Rating Scale (QDRS) | Baseline (Week 0)
  The QDRS is a brief, informant-based tool designed to assess cognitive function and detect dementia quickly, typically in 3-5 minutes. It evaluates 10 domains, including memory, orientation, decision-making, and daily activities, with scores ranging from 0 to 30, where higher scores indicate greater impairment.
  * 0-1.5: No dementia
  * 2.0-5.5: Mild cognitive impairment (MCI)
  * 6.0-12.5: Mild dementia
  * 13.0-20.5: Moderate dementia
  * 21-30: Severe dementia
Conditioned Pain Modulation (CPM) | Baseline (Week 0) and end of intervention (Week 4).
  Descending pain modulation will be assessed by measuring the change in pressure pain threshold on the trapezius immediately after immersing the contralateral hand up to the wrist in a 12 °C cold-water bath for one minute. An increase in pressure pain threshold following immersion indicates stronger descending pain modulation, with higher CPM scores reflecting better modulation.
Quality of Life Alzheimer's Disease Questionnaire (QOL-AD) | Baseline (Week 0) and end of intervention (Week 4).
  Quality of Life will be assessed using the 13-item QOL-AD, which evaluates physical health, mood, memory, and overall life satisfaction. Each item is rated from 1 (poor) to 4 (excellent), with total scores ranging from 13 to 52; higher scores indicate better QOL. The QOL-AD has high Internal consistency (Cronbach α = 0.80 to 0.89) and strong validity, correlating well with other QOL measures, cognitive function, and mood assessments.
Mini-Montreal Cognitive Assessment (Mini-MoCA) | Pre-baseline screening assessment (prior to Week 0).
  Mini-MoCA: The 5-minute Mini-MoCA is a shortened version of the MoCA, targeting tasks most sensitive to mild cognitive impairment. It takes approximately 5 minutes to administer and assesses five cognitive domains: attention, verbal learning and memory, executive function/language, and orientation. The cut-off score is 12, with 1 point added for persons with less than 12 years of education.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona College of Nursing, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be stored securely electronically via redCAP and physically in locked cabinets within the lab. There is no plan to share IPD with other researchers.

REFERENCES:
- [Background] Zhou Z, Hui ES, Kranz GS, Chang JR, de Luca K, Pinto SM, Chan WW, Yau SY, Chau BK, Samartzis D, Jensen MP, Wong AYL. Potential mechanisms underlying the accelerated cognitive decline in people with chronic low back pain: A scoping review. Ageing Res Rev. 2022 Dec;82:101767. doi: 10.1016/j.arr.2022.101767. Epub 2022 Oct 22. PMID 36280211
- [Background] Thakur ER, Amspoker AB, Sansgiry S, Snow AL, Stanley M, Wilson N, Freshour J, Kunik ME. Pain Among Community-Dwelling Older Adults with Dementia: Factors Associated with Undertreatment. Pain Med. 2017 Aug 1;18(8):1476-1484. doi: 10.1093/pm/pnw225. PMID 27694534
- [Background] Stein C, Clark JD, Oh U, Vasko MR, Wilcox GL, Overland AC, Vanderah TW, Spencer RH. Peripheral mechanisms of pain and analgesia. Brain Res Rev. 2009 Apr;60(1):90-113. doi: 10.1016/j.brainresrev.2008.12.017. Epub 2008 Dec 31. PMID 19150465
- [Background] Sofat N, Smee C, Hermansson M, Howard M, Baker EH, Howe FA, Barrick TR. Functional MRI demonstrates pain perception in hand osteoarthritis has features of central pain processing. J Biomed Graph Comput. 2013 Nov;3(4):10.5430/jbgc.v3n4p20. doi: 10.5430/jbgc.v3n4p20. PMID 24294351
- [Background] Simis M, Reidler JS, Duarte Macea D, Moreno Duarte I, Wang X, Lenkinski R, Petrozza JC, Fregni F. Investigation of central nervous system dysfunction in chronic pelvic pain using magnetic resonance spectroscopy and noninvasive brain stimulation. Pain Pract. 2015 Jun;15(5):423-32. doi: 10.1111/papr.12202. Epub 2014 May 2. PMID 24799153
- [Background] Shen C, Zhao X, Dwibedi N, Wiener RC, Findley PA, Sambamoorthi U. Opioid use and the presence of Alzheimer's disease and related dementias among elderly Medicare beneficiaries diagnosed with chronic pain conditions. Alzheimers Dement (N Y). 2018 Dec 7;4:661-668. doi: 10.1016/j.trci.2018.10.012. eCollection 2018. PMID 30560199
- [Background] Sefat O, Salehinejad MA, Danilewitz M, Shalbaf R, Vila-Rodriguez F. Combined Yoga and Transcranial Direct Current Stimulation Increase Functional Connectivity and Synchronization in the Frontal Areas. Brain Topogr. 2022 Mar;35(2):207-218. doi: 10.1007/s10548-022-00887-z. Epub 2022 Jan 29. PMID 35092544
- [Background] Patel KV, Guralnik JM, Dansie EJ, Turk DC. Prevalence and impact of pain among older adults in the United States: findings from the 2011 National Health and Aging Trends Study. Pain. 2013 Dec;154(12):2649-2657. doi: 10.1016/j.pain.2013.07.029. PMID 24287107
- [Background] Parks EL, Geha PY, Baliki MN, Katz J, Schnitzer TJ, Apkarian AV. Brain activity for chronic knee osteoarthritis: dissociating evoked pain from spontaneous pain. Eur J Pain. 2011 Sep;15(8):843.e1-14. doi: 10.1016/j.ejpain.2010.12.007. Epub 2011 Feb 10. PMID 21315627
- [Background] Park J, Tolea MI, Sherman D, Rosenfeld A, Arcay V, Lopes Y, Galvin JE. Feasibility of Conducting Nonpharmacological Interventions to Manage Dementia Symptoms in Community-Dwelling Older Adults: A Cluster Randomized Controlled Trial. Am J Alzheimers Dis Other Demen. 2020 Jan-Dec;35:1533317519872635. doi: 10.1177/1533317519872635. Epub 2019 Sep 18. PMID 31533443
- [Background] Park J, Sherman DG, Agogo G, Hoogendijk EO, Liu Z. Frailty modifies the intervention effect of chair yoga on pain among older adults with lower extremity osteoarthritis: Secondary analysis of a nonpharmacological intervention trial. Exp Gerontol. 2020 Jun;134:110886. doi: 10.1016/j.exger.2020.110886. Epub 2020 Feb 20. PMID 32088398
- [Background] Park J, McCaffrey R, Newman D, Cheung C, Hagen D. The effect of Sit 'n' Fit Chair Yoga among community-dwelling older adults with osteoarthritis. Holist Nurs Pract. 2014 Jul-Aug;28(4):247-57. doi: 10.1097/HNP.0000000000000034. PMID 24919095
- [Background] Park J, McCaffrey R, Dunn D, Goodman R. Managing osteoarthritis: comparisons of chair yoga, Reiki, and education (pilot study). Holist Nurs Pract. 2011 Nov-Dec;25(6):316-26. doi: 10.1097/HNP.0b013e318232c5f9. PMID 22015342
- [Background] Park J, Hung L, Randhawa P, Surage J, Sullivan M, Levine H, Ortega M. 'Now I can bend and meet people virtually in my home': The experience of a remotely supervised online chair yoga intervention and visual socialisation among older adults with dementia. Int J Older People Nurs. 2023 Jan;18(1):e12513. doi: 10.1111/opn.12513. Epub 2022 Nov 14. PMID 36373431
- [Background] Park J, Heilman KJ, Sullivan M, Surage J, Levine H, Hung L, Ortega M, Kirk Wiese LA, Ahn H. Remotely supervised home-based online chair yoga intervention for older adults with dementia: Feasibility study. Complement Ther Clin Pract. 2022 Aug;48:101617. doi: 10.1016/j.ctcp.2022.101617. Epub 2022 Jun 14. PMID 35738115
- [Background] Martorella G, Miao H, Wang D, Park L, Mathis K, Park J, Sheffler J, Granville L, Teixeira AL, Schulz PE, Ahn H. Feasibility, Acceptability, and Efficacy of Home-Based Transcranial Direct Current Stimulation on Pain in Older Adults with Alzheimer's Disease and Related Dementias: A Randomized Sham-Controlled Pilot Clinical Trial. J Clin Med. 2023 Jan 4;12(2):401. doi: 10.3390/jcm12020401. PMID 36675330
- [Background] Luedtke K, Rushton A, Wright C, Jurgens T, Polzer A, Mueller G, May A. Effectiveness of transcranial direct current stimulation preceding cognitive behavioural management for chronic low back pain: sham controlled double blinded randomised controlled trial. BMJ. 2015 Apr 16;350:h1640. doi: 10.1136/bmj.h1640. PMID 25883244
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Hiramatsu T, Nakanishi K, Yoshimura S, Yoshino A, Adachi N, Okamoto Y, Yamawaki S, Ochi M. The dorsolateral prefrontal network is involved in pain perception in knee osteoarthritis patients. Neurosci Lett. 2014 Oct 3;581:109-14. doi: 10.1016/j.neulet.2014.08.027. Epub 2014 Aug 26. PMID 25168605
- [Background] Gwilym SE, Keltner JR, Warnaby CE, Carr AJ, Chizh B, Chessell I, Tracey I. Psychophysical and functional imaging evidence supporting the presence of central sensitization in a cohort of osteoarthritis patients. Arthritis Rheum. 2009 Sep 15;61(9):1226-34. doi: 10.1002/art.24837. PMID 19714588
- [Background] Fregni F, Nitsche MA, Loo CK, Brunoni AR, Marangolo P, Leite J, Carvalho S, Bolognini N, Caumo W, Paik NJ, Simis M, Ueda K, Ekhitari H, Luu P, Tucker DM, Tyler WJ, Brunelin J, Datta A, Juan CH, Venkatasubramanian G, Boggio PS, Bikson M. Regulatory Considerations for the Clinical and Research Use of Transcranial Direct Current Stimulation (tDCS): review and recommendations from an expert panel. Clin Res Regul Aff. 2015 Mar 1;32(1):22-35. doi: 10.3109/10601333.2015.980944. PMID 25983531
- [Background] Danilewitz M, Gao S, Salehinejad MA, Ge R, Nitsche MA, Vila-Rodriguez F. Effect of combined yoga and transcranial direct current stimulation intervention on working memory and mindfulness. J Integr Neurosci. 2021 Jun 30;20(2):367-374. doi: 10.31083/j.jin2002036. PMID 34258935
- [Background] Better, M. A. (2023). Alzheimer's disease facts and figures. Alzheimers Dement, 19(4), 1598-1695. Center for Disease Control and Prevention. (2024). National Insitutes of Health. www.cdc.gov Chen, J., Wang, X., & Xu, Z. (2023). The Relationship Between Chronic Pain and Cognitive Impairment in the Elderly: A Review of Current Evidence. J Pain Res, 16, 2309-2319. https://doi.org/10.2147/jpr.S416253
- [Background] Antal A, Terney D, Kuhnl S, Paulus W. Anodal transcranial direct current stimulation of the motor cortex ameliorates chronic pain and reduces short intracortical inhibition. J Pain Symptom Manage. 2010 May;39(5):890-903. doi: 10.1016/j.jpainsymman.2009.09.023. PMID 20471549
- [Background] Ahn H, Zhong C, Miao H, Chaoul A, Park L, Yen IH, Vila MA, Sorkpor S, Abdi S. Efficacy of combining home-based transcranial direct current stimulation with mindfulness-based meditation for pain in older adults with knee osteoarthritis: A randomized controlled pilot study. J Clin Neurosci. 2019 Dec;70:140-145. doi: 10.1016/j.jocn.2019.08.047. Epub 2019 Aug 14. PMID 31421990
- [Background] Ahn H, Woods AJ, Kunik ME, Bhattacharjee A, Chen Z, Choi E, Fillingim RB. Efficacy of transcranial direct current stimulation over primary motor cortex (anode) and contralateral supraorbital area (cathode) on clinical pain severity and mobility performance in persons with knee osteoarthritis: An experimenter- and participant-blinded, randomized, sham-controlled pilot clinical study. Brain Stimul. 2017 Sep-Oct;10(5):902-909. doi: 10.1016/j.brs.2017.05.007. Epub 2017 May 19. PMID 28566193
- [Background] Ahn H, W. A., Choi E, Padhye N, Fillingim R. (2017). Efficacy of transcranial direct current stimulation on clinical pain severity in older adults with knee osteoarthritis pain: A double-blind, randomized, sham-controlled pilot clinical study. Journal of Pain, 18(4), S87-S88.
- [Background] Ahn H, Suchting R, Woods AJ, Miao H, Green C, Cho RY, Choi E, Fillingim RB. Bayesian analysis of the effect of transcranial direct current stimulation on experimental pain sensitivity in older adults with knee osteoarthritis: randomized sham-controlled pilot clinical study. J Pain Res. 2018 Sep 27;11:2071-2082. doi: 10.2147/JPR.S173080. eCollection 2018. PMID 30310309
- [Background] Ahn H, Sorkpor S, Miao H, Zhong C, Jorge R, Park L, Abdi S, Cho RY. Home-based self-administered transcranial direct current stimulation in older adults with knee osteoarthritis pain: An open-label study. J Clin Neurosci. 2019 Aug;66:61-65. doi: 10.1016/j.jocn.2019.05.023. Epub 2019 May 29. PMID 31153751
- [Background] Ahn H, Galle K, Mathis KB, Miao H, Montero-Hernandez S, Jackson N, Ju HH, McCrackin H, Goodwin C, Hargraves A, Jain B, Dinh H, Abdul-Mooti S, Park L, Pollonini L. Feasibility and efficacy of remotely supervised cranial electrical stimulation for pain in older adults with knee osteoarthritis: A randomized controlled pilot study. J Clin Neurosci. 2020 Jul;77:128-133. doi: 10.1016/j.jocn.2020.05.003. Epub 2020 May 8. PMID 32402609